CLINICAL TRIAL: NCT03017898
Title: Treatment of Anal Fistula With Laser Mediated Heat Coagulation Using Fistula Laser Closure (FiLaC)
Brief Title: Treatment of Anal Fistula With Lasercoagulation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted due to lower success rates than expected, under evaluation, will potentially resume at a later date.
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FiLaC-2016
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Fistula-In-Ano; Anal Fistula
Keywords: FiLaC; Fistula Laser Closure; Laser Coagulation
MeSH Terms: conditions — Rectal Fistula | interventions — Laser Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser coagulation (Experimental): Treatment of anal fistulae meeting the inclusion criteria
  Interventions: Procedure: Laser Coagulation

INTERVENTIONS:
Procedure: Laser Coagulation — Laser coagulation of anal fistula
  Other Names: Fistula Laser Closure (FiLaC)

SUMMARY:
The purpose of this study is to determine whether treatment with laser coagulation is an effective and safe treatment option for patients with anal fistula

DETAILED DESCRIPTION:
Treatment of anal fistula remains a challenge - the only truly effective treatment available (fistulotomy) involves very high rates of anal incontinence if performed on the majority of patients, and a vast number of alternative, sphincter-preserving treatments have been developed and evaluated in the past decades. The treatment of anal fistula with laser coagulation causes the fistula to collapse and subsequently heal, without having to add any external materials. The available published studies show that the treatment is safe regarding infection and incontinence, and that a majority of the patients treated show complete healing. There is however a need for more prospective studies to ascertain these preliminary facts.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.
2. Subject must be at least 18 years of age
3. Subject must have a verified anal fistula (by transanal ultrasound performed by treating surgeon)
4. Subject must have a clean and infection-free fistula tract (no cavities seen on transanal ultrasound)
5. Subject must be able to comply with study and study follow-up requirements.

Exclusion Criteria:

1. Subject with anorectal fistula due to Crohn's disease
2. Subject has an undrained abscess in fistula tract (cavities as seen on transanal ultrasound)
3. Subject has fistula with side tracts (as seen on transanal ultrasound)
4. Subject is unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Healing | 12 months
  Fistula closure success at 12 months is defined as complete healing of the fistula tract and external opening at clinical examination and on a transanal ultrasound performed by the examining surgeon (yes/no).

SECONDARY OUTCOMES:
Infection | 12 months
  Rate of infection i.e. formation of abcess during the time of healing or thereafter within the first year of treatment.
Incontinence | 12 months
  Presence of fecal incontinence as described by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilhelm A. A new technique for sphincter-preserving anal fistula repair using a novel radial emitting laser probe. Tech Coloproctol. 2011 Dec;15(4):445-9. doi: 10.1007/s10151-011-0726-0. Epub 2011 Aug 16. PMID 21845480
- [Background] Giamundo P, Esercizio L, Geraci M, Tibaldi L, Valente M. Fistula-tract Laser Closure (FiLaC): long-term results and new operative strategies. Tech Coloproctol. 2015 Aug;19(8):449-53. doi: 10.1007/s10151-015-1282-9. Epub 2015 Feb 28. PMID 25724967
- [Background] Giamundo P, Geraci M, Tibaldi L, Valente M. Closure of fistula-in-ano with laser--FiLaC: an effective novel sphincter-saving procedure for complex disease. Colorectal Dis. 2014 Feb;16(2):110-5. doi: 10.1111/codi.12440. PMID 24119103
- [Background] Ozturk E, Gulcu B. Laser ablation of fistula tract: a sphincter-preserving method for treating fistula-in-ano. Dis Colon Rectum. 2014 Mar;57(3):360-4. doi: 10.1097/DCR.0000000000000067. PMID 24509460